CLINICAL TRIAL: NCT00389389
Title: A Phase I, Open-Label, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD4877 Administered Weekly or Every Two Weeks in Patients With Advanced Solid Malignancies
Brief Title: Phase I, Open-Label, Dose-Escalation Study of AZD4877 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2782C00001
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2009-05-01 (Estimated); Status verified 2009-04

CONDITIONS: Neoplasms
Keywords: Advanced Solid Malignancies; Advanced solid tumors; Cancer; Phase I; Solid tumors; Solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — N-(3-aminopropyl)-N-(1-(5-benzyl-3-methyl-4-oxo-(1,2)thiazolo(5,4-d)pyrimidin-6-yl)-2-methylpropyl)-4-methylbenzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AZD4877 — intravenous infusion

SUMMARY:
The primary purpose of this study is to find out what the maximum tolerated dose is for an experimental drug called AZD4877 based on the side effects experiences by patients that receive AZD4877 on a weekly basis

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors for which standard treatment doesn't exist or is no longer effective.
* Relatively good overall health other than your cancer.

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells).
* Serious heart conditions.
* Poor liver or kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To identify a maximum-tolerated dose of AZD4877 by assessment of the incidence of dose-limiting toxicities as measured by the Common Terminology Criteria for Adverse Events (CTCAE) grade and type of AEs experienced in the first cycle of treatment. | assessed at each treatment

SECONDARY OUTCOMES:
Pharmacokinetics parameters of Cmax, AUC and C24 of AZD4877 measured during the first cycle of treatment. | Assessed after the first course of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ochs, MD, Study Director — AstraZeneca
Locations (3):
- United States (3):
  - Research Site, Denver, Colorado
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas